CLINICAL TRIAL: NCT00518986
Title: Double-Blind, Placebo-Controlled, Study to Evaluate the Efficacy and Safety of Armodafinil for Adults With Excessive Sleepiness Associated With Obstructive Sleep Apnea/Hypopnea Syndrome With Major Depressive Disorder or Dysthymic Disorder
Brief Title: Efficacy and Safety of Armodafinil for Adults With Excessive Sleepiness Obstructive Sleep Apnea/Hypopnea and Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/4024/ES/US
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Results first posted 2011-03-29 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Sleep Disorders; Obstructive Sleep Apnea; Major Depressive Disorder; Dysthymic Disorder
Keywords: Obstructive Sleep Apnea/Hypopnea Syndrome; Excessive Sleepiness
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea, Obstructive; Depressive Disorder, Major; Dysthymic Disorder; Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): armodafinil 200 mg/day
  Interventions: Drug: armodafinil
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: armodafinil — 200 mg/day
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The primary objective of the study is to evaluate whether armodafinil at a target dosage of 200 mg/day is more effective than placebo treatment in improving excessive sleepiness in patients with obstructive sleep apnea/hypopnea syndrome (OSAHS) who have comorbid major depressive disorder or dysthymic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of obstructive sleep apnea/hypopnea syndrome (OSAHS)
* Complaint of residual excessive sleepiness despite nasal continuous positive airway pressure (nCPAP) therapy being effective
* Current or prior diagnosis of major depressive disorder or dysthymic disorder
* Clinically stable with regard to depressed mood and has shown a treatment response to selective serotonin reuptake inhibitor (SSRI) therapy or serotonin and norepinephrine reuptake inhibitor (SNRI) therapy
* Patient has been on a stable monotherapy dose of an allowed SSRI or SNRI for at least 8 weeks at the time of screening
* Women of childbearing potential must use a medically accepted method of contraception.

Exclusion Criteria:

* Confirmed or suspected diagnosis of a currently active sleep disorder other than obstructive sleep apnea/hypopnea syndrome (OSAHS)
* Current episode of major depression that is considered to be treatment-resistant
* A primary diagnosis of: eating disorder, psychotic disorder, delirium, dementia, substance-related disorders, or moderate to severe hypochondriasis
* Patient has a history of bipolar disorder, psychotic depression, schizophrenia, schizoaffective disorder, any other psychotic disorder, or other clinically significant uncontrolled psychiatric condition.
* Patient has a history of homicidal ideation or significant aggression
* Patient has a diagnosis of severe antisocial or borderline personality disorder
* Has a history of significant suicidal ideation, or has current active suicidal ideation, or is considered at imminent risk of self harm.
* Patient has a history consistent with fibromyalgia or chronic fatigue syndrome
* A high consumption of caffeinated products, approximately equivalent to 5 or more cups of coffee per day
* Patient history of any clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction
* Has a past or present seizure disorder
* Patient has a history of alcohol, narcotic, or any other substance abuse or dependence (with the exception of nicotine)
* Psychotherapeutic intervention for the patient was initiated within 8 weeks of the screening visit.
* Patient has known human immunodeficiency virus (HIV)
* Patient has any clinically significant uncontrolled medical condition (including illnesses related to the cardiovascular, renal, or hepatic systems) or surgical condition (treated or untreated)
* Patient is a pregnant or lactating woman
* Patient has previously received armodafinil; or, patient has used modafinil or any investigational product within 28 days of the baseline visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Pulmonary Associates, P.A., Phoenix, Arizona
  - Psypharma Clinical Research, Phoenix, Arizona
  - PsyPharm Clinical Research, Inc., Tucson, Arizona
  - Behavioral Research Specialists, Glendale, California
  - California Clinical Trials Medical Group, Inc., Glendale, California
  - Pacific Sleep Medicine Services, Inc., Redlands, California
  - Pacific Research Network, Inc., San Diego, California
  - Pacific Sleep Medicine Services, Inc., San Diego, California
  - California Clinical Trials Medical Group, Inc., San Diego, California
  - SDS Clinical Research, Santa Ana, California
  - St. Johns Medical Plaza Sleep Disorders Center, Santa Monica, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - PAB Clinical Research, Brandon, Florida
  - Florida Sleep Institute, Spring Hill, Florida
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - SomnoMedics, Tampa, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Florida Pulmonary Research Center, LLC, Winter Park, Florida
  - The Sleep Disorders Center, Atlanta, Georgia
  - Neurotrials Research, Inc, Atlanta, Georgia
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - SleepMed, Inc, Macon, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Peoria Pulmonary Associates, Peoria, Illinois
  - Sleep and Behavior Medicine, Vernon Hills, Illinois
  - The Center for Sleep and Wake Disorders, Danville, Indiana
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Community Research, Crestview, Kentucky
  - Clinical Trials of America, Shreveport, Louisiana
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Sleep Health Centers, Brighton, Massachusetts
  - AccelRx Research, Fall River, Massachusetts
  - The Center for Sleep Medicine, Hattiesburg, Mississippi
  - Washington University, St Louis, Missouri
  - Somnos Sleep Center, Lincoln, Nebraska
  - Brooklyn Medical Institute, Brooklyn, New York
  - Clinilabs, Inc, New York, New York
  - Sleep Medicine Centers, West Seneca, New York
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Trials of America, Hickory, North Carolina
  - Tri-State Sleep Disorders Center, Cincinnati, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sleep Lab of Northeastern PA, Clarks Summit, Pennsylvania
  - University of Pennsylvania Center for Sleep, Philadelphia, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - University Services, West Chester, Pennsylvania
  - AccelRx Research, Lincoln, Rhode Island
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - SleepMed of South Carolina, Columbia, South Carolina
  - Sleep Medicine of Middle Tennessee, Nashville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Sleep Medicine Associates of Texas, P.A., Dallas, Texas
  - Baylor College of Medicine VAMC Sleep Research, Houston, Texas
  - Houston Sleep Center, Houston, Texas
  - Northwest Clinical Research, Bellevue, Washington
  - Pacific Sleep Medicine Services, Inc., Seattle, Washington

REFERENCES:
- [Derived] Krystal AD, Harsh JR, Yang R, Rippon GA, Lankford DA. A double-blind, placebo-controlled study of armodafinil for excessive sleepiness in patients with treated obstructive sleep apnea and comorbid depression. J Clin Psychiatry. 2010 Jan;71(1):32-40. doi: 10.4088/JCP.09m05536gry. Epub 2009 Dec 29. PMID 20051221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 centers in the US. First participant enrolled: October 2007/ Last participant last visit: March 2009
Pre-assignment Details: The study consisted of a 1-week single-blind, placebo run-in screening period followed by a 12-week double blind treatment period. Of the 249 patients enrolled, 248 patients received at least 1 dose of study drug and were evaluated for safety; 1 patient who was assigned to receive armodafinil was lost to follow-up before taking any study drug.
Groups:
- Armodafinil 200 mg/Day: Armodafinil (or placebo) was titrated to a target dosage of 200 mg/day (4 tablets) for each patient. Dosing began at 50 mg (1 tablet)/day each morning on Day 1, and then increased by 50 mg (1 tablet) on days 2, 5, and 8 to target dose of 200 mg/day (4 tablets). If deemed appropriate by investigator, dose could be further titrated to 250 mg/day (5 tablets). If tolerability issues arose, dose could be decreased in 50 mg increments anytime after 200 mg/day dose was achieved.
- Placebo: Placebo tablets matching the 50 mg armodafinil tablet were used in a manner identical to that of the armodafinil tablets for both the placebo run in period and the double blind treatment period. Study drug was titrated to a target dosage of 4 tablets/day for each patient. Dosing began at 1 tablet/day in the morning on Day 1, and then increased by 1 tablet on days 2, 5, and 8 to target dose of 4 tablets. If deemed appropriate by investigator, dose could be further titrated to 5 tablets. If tolerability issues arose, dose could be decreased in 1 tablet increments anytime after 4 tablets/day dose was achieved.
Period: Overall Study
Arm/Group | Armodafinil 200 mg/Day | Placebo
Started | 125 (One subject discontinued before treatment, only 124 subjects in each treatment group were dosed.) | 124
Completed | 99 | 98
Not Completed | 26 | 26
Not completed — Adverse Event | 12 | 7
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 5 | 7
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Non-Specific | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil 200 mg/Day | Placebo | Total
Number analyzed (Participants) | 125 | 124 | 249
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 124 | 249
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.5 (10.32) | 49.5 (9.69) | 49.5 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 66 | 134
  Male | 57 | 58 | 115
Region of Enrollment [Number; unit: participants]
  United States | 125 | 124 | 249

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Maintenance of Wakefulness Test (MWT) to Endpoint (12 Weeks or Last Observation After Baseline)
Description: MWT measures ability of subject to remain awake. Subjects instructed to try and remain awake during series of 4 30-minute periods (0900, 1100, 1300, and 1500) reclining in dark room. Each period was terminated immediately after sleep onset or at end of 30 minutes if no sleep occurred. If subject fell asleep, they were awakened and not allowed to sleep for remainder of that 30 minute period. Change from Baseline to Endpoint (12 weeks or last observation after baseline) in mean sleep latency averaged from the 4 intervals was measured. Poorest outcome was 0 minutes the best was 30 minutes.
Time Frame: Baseline and 12 weeks (or last observation after baseline)
Population: Full analysis set which includes subjects who had at least 1 measurement of MWT or Clinical Global Impression of Change (CGI-C) after baseline.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 109 | 105
Minutes | 2.6 (7.09) | 1.1 (7.61)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Since there were two primary outcome measures the Hochberg procedure was used to control overall Type 1 error rate at the 0.05 level. If both p-values for the primary variables were <= 0.05 the treatment was claimed to be significant for both variables. If 1 p-value was > 0.05and the other was <=0.025, the variable with a p-value <= 0.025 was claimed as significant; Test type: Superiority or Other; p = 0.3043, ANCOVA; Study drug was fixed factor and corresponding baseline value was a covariate

2. Primary Outcome: Clinical Global Impression of Change (CGI-C) at Endpoint (12-weeks or Last Observation After Baseline)
Description: The CGI-C is a clinician's rating of disease severity compared with baseline as assessed by Clinical Global Impression of Severity (CGI-S). CGI-C rates improvement by 7 categories: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. CGI-S measured 7 categories of illness as well: normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among most extremely ill. Proportion of responders who had at least "minimally improved" in CGI-C ratings (as related to sleepiness) were assessed.
Time Frame: 12 weeks (or last observation after baseline)
Population: Full analysis set which includes subjects who had at least 1 measurement of MWT or CGI-C after baseline.
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 113 | 112
Participants
  At least minimal improvement | 78 | 59
  No improvement | 35 | 53
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0120, Chi-squared; P-value for comparison is from a Pearson's chi-square test

3. Secondary Outcome: Change From Baseline on the Epworth Sleepiness Scale (ESS) at Endpoint (12 Weeks or Last Measurement After Baseline)
Description: For this key secondary outcome the ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The change in ESS total score from baseline to Endpoint (12 weeks or last observation after baseline) are summarized.
Time Frame: Baseline and 12 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who had at least one assessment of ESS after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 113 | 112
Units on a scale | -6.5 (0.44) | -4.6 (0.44)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Least squares (LS) mean and standard error of the LS mean for each treatment group, and p-value for the treatment comparison is from an analysis of covariance (ANCOVA) with treatment as a factor and the baseline as covariate; Test type: Superiority or Other; p = 0.0027, ANCOVA — Nominal p-value is presented, but statistical significance cannot be claimed. As a key secondary variable significance could be claimed only if treatment effect was significant for both primary efficacy variables

4. Secondary Outcome: Change From Baseline on Maintenance of Wakefulness Test (MWT) at 4 Weeks
Description: MWT measures ability of subject to remain awake. Subjects instructed to try and remain awake during series of four 30-minute periods (0900, 1100, 1300, and 1500) reclining in dark room. Each period was terminated immediately after sleep onset or at end of 30 minutes if no sleep occured. If subject fell asleep, they were awakened and not allowed to sleep for remainder of that 30 minute period. Change from Baseline to 4 weeks in mean sleep latency (measured in minutes)averaged from each of the four testing intervals was measured. The poorest outcome was 0 minutes the best was 30 minutes.
Time Frame: baseline and 4 weeks
Population: Full analysis set defined as subjects who had MWT measurement at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 108 | 105
Minutes | 2.7 (0.63) | -0.1 (0.64)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0019, ANCOVA

5. Secondary Outcome: Change From Baseline on Maintenance of Wakefulness Test (MWT) at 8 Weeks
Description: MWT measures ability of subject to remain awake. Subjects instructed to try and remain awake during series of four 30-minute periods (0900, 1100, 1300, and 1500) reclining in dark room. Each period was terminated immediately after sleep onset or at end of 30 minutes if no sleep occured. If subject fell asleep, they were awakened and not allowed to sleep for remainder of that 30 minute period. Change from Baseline to 8 weeks in mean sleep latency (measured in minutes)averaged from each of the four testing intervals was measured. The poorest outcome was 0 minutes the best was 30 minutes.
Time Frame: Baseline and 8 weeks following start of study drug administration
Population: Full analysis set defined as subjects with MWT measure at 8 weeks and baseline
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 100
Minutes | 2.1 (0.61) | 1.2 (0.62)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.3145, ANCOVA

6. Secondary Outcome: Change From Baseline on Maintenance of Wakefulness Test (MWT) at 12 Weeks
Description: MWT measures ability of subject to remain awake. Subjects instructed to try and remain awake during series of four 30-minute periods (0900, 1100, 1300, and 1500) reclining in dark room. Each period was terminated immediately after sleep onset or at end of 30 minutes if no sleep occured. If subject fell asleep, they were awakened and not allowed to sleep for remainder of that 30 minute period. Change from Baseline to 12 weeks in mean sleep latency (measured in minutes)averaged from each of the four testing intervals was measured. The poorest outcome was 0 minutes the best was 30 minutes.
Time Frame: baseline and 12 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who had measurements of MWT at baseline and 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 96 | 95
Minutes | 2.5 (0.64) | 1.4 (0.64)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.2196, ANCOVA

7. Secondary Outcome: Clinical Global Impression of Change (CGI-C) at 4 Weeks
Description: The CGI-C is a clinician's rating of disease severity compared with baseline as assessed by Clinical Global Impression of Severity (CGI-S). CGI-C rates 7 responses: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. CGI-S measured 7 categories as well: normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among most extremely ill. Proportion of responders who had at least "minimally improved" in CGI-C ratings (as related to sleepiness) at 4 weeks were assessed.
Time Frame: 4 weeks after beginning study drug treatment
Population: Full analysis set defined as subjects who were assessed with CGI-C at 4 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 111 | 108
Participants
  At least minimal improvement | 75 | 64
  No improvement | 36 | 44
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.2017, Chi-squared — P-value is from Pearson's chi-square test

8. Secondary Outcome: Clinical Global Impression of Change (CGI-C) at 8 Weeks
Description: The CGI-C is a clinician's rating of disease severity compared with baseline as assessed by Clinical Global Impression of Severity (CGI-S). CGI-C rates 7 responses: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. CGI-S measured 7 categories as well: normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among most extremely ill. Proportion of responders who had at least "minimally improved" in CGI-C ratings (as related to sleepiness) at 8 weeks were assessed.
Time Frame: 8 weeks after beginning study drug treatment
Population: Full analysis set defined as subjects assessed by CGI-C at 8 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 98
Participants
  At least minimal improvement | 76 | 52
  No improvement | 28 | 46
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0032, Chi-squared — P-value from Pearson's chi-square test

9. Secondary Outcome: Clinical Global Impression of Change (CGI-C) at 12 Weeks
Description: The CGI-C is a clinician's rating of disease severity compared with baseline as assessed by Clinical Global Impression of Severity (CGI-S). CGI-C rates 7 responses: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. CGI-S measured 7 categories as well: normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among most extremely ill. Proportion of responders who had at least minimal improvement in CGI-C ratings (as related to sleepiness) were assessed.
Time Frame: 12 weeks after beginning treatment
Population: Full analysis set defined as subjects assessed with CGI-C at week 12
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 96 | 95
Participants
  At least minimal improvement | 69 | 53
  No improvement | 27 | 42
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0207, Chi-squared — P-value from Pearson's chi-square test

10. Secondary Outcome: Clinical Global Impression of Change (CGI C) at 4 Weeks - Full Scale
Description: The CGI-C is a clinician's rating of disease severity compared with baseline as assessed by Clinical Global Impression of Severity (CGI-S). CGI-C rates 7 responses: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. CGI-S measured 7 categories as well: normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among most extremely ill. The results for the number of participants who responded to each item on the full scale at 4 weeks are presented.
Time Frame: 4 weeks after start of treatment
Population: Full analysis set defined as subjects who were assessed by CGI-C at 4 weeks.
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 111 | 108
Participants
  Very much improved | 15 | 11
  Much improved | 34 | 21
  Minimally improved | 26 | 32
  No change | 32 | 37
  Minimally worse | 3 | 5
  Much worse | 1 | 2
  Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0529, Cochran-Mantel-Haenszel — P-value was generated from a Cochran-Mantel-Haenszel chi-square test

11. Secondary Outcome: Clinical Global Impression of Change (CGI-C) at 8 Weeks - Full Scale
Description: The CGI-C is a clinician's rating of disease severity compared with baseline as assessed by Clinical Global Impression of Severity (CGI-S). CGI-C rates 7 responses: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. CGI-S measured 7 categories as well: normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among most extremely ill. The results for the number of participants who responded to each item on the full scale at 8 weeks are presented.
Time Frame: 8 weeks after start of study drug treatment
Population: Full analysis set defined as subjects who were assessed by CGI-C at 8 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 98
Participants
  Very much improved | 16 | 11
  Much improved | 39 | 19
  Minimally improved | 21 | 22
  No change | 26 | 37
  Minimally worse | 1 | 7
  Much worse | 1 | 2
  Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel

12. Secondary Outcome: Clinical Global Impression of Change (CGI-C) at 12 Weeks - Full Scale
Description: The CGI-C is a clinician's rating of disease severity compared with baseline as assessed by Clinical Global Impression of Severity (CGI-S). CGI-C rates 7 responses: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. CGI-S measured 7 categories as well: normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among most extremely ill. The results for the number of participants who responded to each item on the full scale at 12 weeks are presented.
Time Frame: 12 weeks after starting study drug treatment
Population: Full analysis set defined as subjects assessed by CGI-C at 12 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 96 | 95
Participants
  Very much improved | 27 | 11
  Much improved | 20 | 22
  Minimally improved | 22 | 20
  No change | 22 | 34
  Minimally worse | 4 | 7
  Much worse | 1 | 1
  Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0064, Cochran-Mantel-Haenszel

13. Secondary Outcome: Change From Baseline on Epworth Sleepiness Scale (ESS) at 2 Weeks
Description: ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The change in ESS total score from baseline to two weeks are summarized.
Time Frame: Baseline and 2 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the ESS at baseline and at 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 107 | 104
Unit on a scale | -4.8 (0.40) | -3.8 (0.40)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Least square (LS) mean and standard error of the LS mean for each treatment group, and the p-value for the treatment comparison is from an analysis of covariance (ANCOVA) with treatment as a factor and the baseline value as a covariate; Test type: Superiority or Other; p = 0.1072, ANCOVA

14. Secondary Outcome: Change From Baseline on Epworth Sleepiness Scale (ESS) at 4 Weeks
Description: ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The change in ESS total score from baseline to 4 weeks are summarized.
Time Frame: Baseline and 4 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed ESS at baseline and at Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 111 | 108
Units on a scale | -5.5 (0.42) | -4.2 (0.43)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0355, ANCOVA

15. Secondary Outcome: Change From Baseline on Epworth Sleepiness Scale (ESS) at 8 Weeks
Description: ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The change in ESS total score from baseline to 8 weeks are summarized.
Time Frame: Baseline and 8 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed ESS at Baseline and at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 103 | 98
Units on a scale | -6.0 (0.44) | -4.8 (0.45)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0591, ANCOVA

16. Secondary Outcome: Change From Baseline on Epworth Sleepiness Scale (ESS) at 12 Weeks
Description: ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The change in ESS total score from baseline to 12 weeks are summarized.
Time Frame: 12 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who completed ESS at Baseline and at 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 96 | 95
Units on a scale | -6.8 (0.48) | -4.8 (0.48)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0025, ANCOVA

17. Secondary Outcome: Number of Responders According to the Epworth Sleepiness Scale (ESS) Total Score at 2 Weeks
Description: ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The number of responders who had a total ESS score < 10 and the number of non-responders with a total score >= 10 at 2 weeks are presented.
Time Frame: 2 weeks
Population: Full analysis set defined as the number of subjects who completed the ESS at 2 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 107 | 104
Participants
  Responders | 54 | 40
  Non-responders | 53 | 64
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0794, Chi-squared — P-value for treatment comparison is from Pearson's chi-square test

18. Secondary Outcome: Number of Responders According to the Epworth Sleepiness Scale (ESS) Total Score at 4 Weeks
Description: ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The number of responders who had a total ESS score < 10 and the number of non-responders with a total score >= 10 at 4 weeks are presented.
Time Frame: 4 weeks
Population: Full analysis set defined as number of subjects who completed ESS at 4 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 111 | 108
Participants
  Responders | 59 | 45
  Non-responders | 52 | 63
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0888, Chi-squared — P-value for the treatment comparison is from a Pearson's chi-square test

19. Secondary Outcome: Number of Responders According to the Epworth Sleepiness Scale (ESS) Total Score at 8 Weeks
Description: ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The number of responders who had a total ESS score < 10 and the number of non-responders with a total score >= 10 at 8 weeks are presented.
Time Frame: 8 weeks
Population: Full analysis set defined as subjects who completed ESS at 8 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 103 | 98
Participants
  Responders | 64 | 47
  Non-responders | 39 | 51
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0433, Chi-squared — P-value for the treatment comparison is from a Pearson's chi-square test

20. Secondary Outcome: Number of Responders According to the Epworth Sleepiness Scale (ESS) Total Score at 12 Weeks
Description: ESS score is based on responses to questions (self administered) that assessed the propensity of the subject to fall asleep in 8 everyday situations (sitting and reading, talking to someone, being stopped in traffic, etc.) Scores for the ESS range from 0 to 24, with a higher score indicating greater daytime sleepiness. The number of responders who had a total ESS score < 10 and the number of non-responders with a total score >= 10 at 12 weeks are presented.
Time Frame: 12 weeks
Population: Full analysis set defined as subjects who completed the ESS at 12 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 96 | 95
Participants
  Responders | 65 | 47
  Non-responders | 31 | 48
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Test type: Superiority or Other; p = 0.0105, Chi-squared — P-value for the treatment comparison is from a Pearson's chi-square test

21. Secondary Outcome: Change From Baseline to Endpoint (Week 12 or Last Observation After Baseline) in the Brief Fatigue Inventory (BFI) Total Score
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The total score is calculated by taking the sum of all 9 rating scales for a minimum score of 0 and a maximum score of 90. This assessment examines the difference in total BFI score from Baseline to 12 weeks or last observation after baseline.
Time Frame: Baseline and 12 weeks following start of study drug administration or last recorded observation
Population: Full analysis set defined as subjects with at least one BFI assessment after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 112 | 110
Units on a scale | -8.9 (1.82) | -3.8 (1.84)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0523, ANCOVA

22. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Total Score at 2 Weeks
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The total score is calculated by taking the sum of all 9 rating scales for a minimum score of 0 and a maximum score of 90. This assessment examines the difference in total BFI score from Baseline to 2 weeks.
Time Frame: Baseline and 2 weeks after start of study drug administration
Population: Full analysis set defined as subjects who had completed BFI at baseline and at 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 110 | 106
Units on a scale | -6.1 (1.67) | -0.9 (1.70)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0289, ANCOVA

23. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Total Score at 4 Weeks
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The total score is calculated by taking the sum of all 9 rating scales for a minimum score of 0 and a maximum score of 90. This assessment examines the difference in total BFI score from Baseline to 4 weeks.
Time Frame: Baseline and 4 weeks after start of study drug administration
Population: Full analysis set defined as subjects who had completed BFI at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 111 | 107
Units on a scale | -9.5 (1.72) | -5.8 (1.75)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.1272, ANCOVA

24. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Total Score at 8 Weeks
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The total score is calculated by taking the sum of all 9 rating scales for a minimum score of 0 and a maximum score of 90. This assessment examines the difference in total BFI score from Baseline to 8 weeks.
Time Frame: Baseline and 8 weeks after start of study drug administration
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 97
Units on a scale | -8.8 (1.90) | -3.0 (1.97)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0349, ANCOVA

25. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Total Score at 12 Weeks
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The total score is calculated by taking the sum of all 9 rating scales for a minimum score of 0 and a maximum score of 90. This assessment examines the difference in total BFI score from Baseline to 12 weeks.
Time Frame: Baseline and 12 weeks after start of study drug administration
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 95 | 94
Units on a scale | -10.5 (1.92) | -3.3 (1.93)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0094, ANCOVA

26. Secondary Outcome: Change From Baseline on the Brief Fatigue Inventory (BFI) Worst Daily Fatigue Score at Endpoint (12 Weeks or Last Observation After Baseline)
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with >= 7 indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. This measure compares the change in score from baseline to Week 12 (or last observation after baseline).
Time Frame: Baseline and 12 weeks or last observation after baseline
Population: Full analysis set defined as subjects with at least one observation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 112 | 110
Units on a scale | -1.3 (0.24) | -0.7 (0.24)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0754, ANCOVA

27. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Worse Daily Fatigue Score at 2 Weeks
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. This measure compares the change in score from baseline to Week 2.
Time Frame: Baseline and 2 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed BFI at baseline and at 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 110 | 107
Units on a scale | -1.1 (0.23) | -0.2 (0.24)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0105, ANCOVA

28. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Worse Daily Fatigue Score at 4 Weeks
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. This measure compares the change in score from baseline to Week 4.
Time Frame: Baseline and 4 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed BFI at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 111 | 107
Units on a scale | -1.2 (0.23) | -0.8 (0.24)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.2888, ANCOVA

29. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Worse Daily Fatigue Score at 8 Weeks
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. This measure compares the change in score from baseline to Week 8.
Time Frame: Baseline and 8 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed the BFI at baseline and at week 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 97
Units on a scale | -1.2 (0.24) | -0.3 (0.25)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0130, ANCOVA

30. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Worse Daily Fatigue Score at 12 Weeks
Description: The Brief Fatigue Inventory (BFI) is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. This measure compares the change in score from baseline to Week 12.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 96 | 94
Units on a scale | -1.4 (0.26) | -0.6 (0.26)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0354, ANCOVA

31. Secondary Outcome: Number of Responders According to Brief Fatigue Inventory (BFI) Worst Fatigue Score at Endpoint (12 Weeks or Last Observation After Baseline)
Description: The Brief Fatigue Inventory (BFI) assesses the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. Subjects were considered responders if the final Worst Fatigue Score was < 7 at Week 12 or last observation after baseline.
Time Frame: 12 weeks after start of study drug administration (or last observation after baseline)
Population: Full analysis set defined as subjects who had at least one observation after baseline
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 112 | 111
Participants
  Responders | 63 | 56
  Non-responders | 49 | 55
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders are subjects with worst fatigue score < 7 after baseline; Test type: Superiority or Other; p = 0.3854, Chi-squared — P-value for the treatment comparison is from a Pearson's chi-square test

32. Secondary Outcome: Number of Responders According to the Brief Fatigue Inventory (BFI) Worst Fatigue Score at 2 Weeks
Description: The Brief Fatigue Inventory (BFI) assesses the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. Subjects were considered responders if the final Worst Fatigue Score was < 7 at Week 2.
Time Frame: 2 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed BFI at 2 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 110 | 108
Participants
  Responders | 62 | 43
  Non-responders | 48 | 65
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders were defined as subjects with worst fatigue score < 7; Test type: Superiority or Other; p = 0.0145, Chi-squared — P-value for the treatment comparison is from Pearson's chi-square test

33. Secondary Outcome: Number of Responders According to the Brief Fatigue Inventory (BFI) Worst Fatigue Score at 4 Weeks
Description: The Brief Fatigue Inventory (BFI) assesses the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. Subjects were considered responders if the final Worst Fatigue Score was < 7 at Week 4.
Time Frame: 4 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed BFI at 4 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 111 | 108
Participants
  Responders | 62 | 57
  Non-responders | 49 | 51
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders were patients with worst fatigue scores < 7; Test type: Superiority or Other; p = 0.6475, Chi-squared — P-value for the treatment comparison is from a Pearson's chi-square test

34. Secondary Outcome: Number of Responders According to the Brief Fatigue Inventory (BFI) Worst Fatigue Score at 8 Weeks
Description: The Brief Fatigue Inventory (BFI) assesses the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. Subjects were considered responders if the final Worst Fatigue Score was < 7 at Week 8.
Time Frame: 8 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed the BFI at 8 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 98
Participants
  Responders | 63 | 42
  Non-responders | 41 | 56
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders are subjects with worst fatigue score < 7; Test type: Superiority or Other; p = 0.0118, Chi-squared — P-value for the treatment comparison is from Pearson's chi-square test

35. Secondary Outcome: Number of Responders According to the Brief Fatigue Inventory (BFI) Worst Fatigue Score at 12 Weeks
Description: The Brief Fatigue Inventory (BFI) assesses the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The worst daily fatigue score reports the outcome of a single item on the BFI that rates the worst fatigue experienced over the day on a scale from 0 to 10 with 0 being no fatigue and 10 being most severe. Subjects were considered responders if the final Worst Fatigue Score was < 7 at Week 12.
Time Frame: 12 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed the BFI at 12 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 96 | 95
Participants
  Responders | 55 | 48
  Non-responders | 41 | 47
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders are subjects with a worst fatigue score of < 7; Test type: Superiority or Other; p = 0.3483, Chi-squared — P-value for the treatment comparison is from the Pearson's chi-square test

36. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Interference Score at Endpoint (12 Weeks or Last Observation After Baseline)
Description: The Brief Fatigue Inventory (BFI) assesses the impact of fatigue on daily functioning. Simple numeric rating scales from 0 to 10 are used. The higher scores are associated with more severe fatigue, with any score >= 7 considered to be indicative of severe fatigue. The Interference Score consists of 6 questions that ask subjects to rate on a 0 to 10 scale how during the past 24 hours fatigue has interfered with their general activity, mood, walking ability, normal work, relations with other people, and enjoyment of life. The scores are averaged (0-10) for the Interference Score.
Time Frame: Baseline and at endpoint (12 weeks or last observation after baseline)
Population: Full analysis set defined as subjects who had at least one observation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 112 | 110
Units on a scale | -0.9 (0.22) | -0.3 (0.22)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0879, ANCOVA

37. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Interference Score at 2 Weeks
Description: as for outcome 36
Time Frame: Baseline and 2 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed the BFI at baseline and at 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 110 | 107
Units on a scale | -0.6 (0.20) | 0.0 (0.20)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0277, ANCOVA

38. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Interference Score at 4 Weeks
Description: as for outcome 36
Time Frame: Baseline and 4 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed the BFI at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 111 | 107
Units on a scale | -1.0 (0.20) | -0.6 (0.20)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.1245, ANCOVA

39. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Interference Score at 8 Weeks
Description: as for outcome 36
Time Frame: Baseline and 8 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed the BFI at baseline and at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 97
Units on a scale | -0.9 (0.23) | -0.2 (0.23)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0305, ANCOVA

40. Secondary Outcome: Change From Baseline on Brief Fatigue Inventory (BFI) Interference Score at 12 Weeks (or Last Observation After Baseline)
Description: as for outcome 36
Time Frame: Baseline and 12 weeks after start of study drug administration
Population: Full analysis set defined as subjects who completed BFI at baseline and at 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 96 | 94
Units on a scale | -1.1 (0.23) | -0.3 (0.23)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0129, ANCOVA

41. Secondary Outcome: Change From Baseline on Functional Outcomes of Sleep Questionnaire (FOSQ) Total Score at Endpoint (12 Weeks or Last Observation After Baseline)
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum of 2 maximum of 120) was calculated from the responses. The change in total score from baseline to Endpoint (12 weeks or last observation after baseline) is presented here.
Time Frame: Baseline and endpoint (12 weeks after start of study drug or last observation after baseline)
Population: Full analysis set defined as subjects who had at least one observation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 107
Units on a scale | 2.3 (0.26) | 1.5 (0.26)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0308, ANCOVA

42. Secondary Outcome: Change From Baseline on Functional Outcomes of Sleep Questionnaire (FOSQ) Total Score at 2 Weeks
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum = 2 maximum = 120) was calculated from the responses. The change in total score from baseline to 2 weeks is presented here.
Time Frame: baseline and 2 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed FOSQ at baseline and at 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 100 | 103
Units on a scale | 1.7 (0.24) | 1.1 (0.24)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0679, ANCOVA

43. Secondary Outcome: Change From Baseline on Functional Outcomes of Sleep Questionnaire (FOSQ) Total Score at 4 Weeks
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum = 2 maximum = 120) was calculated from the responses. The change in total score from baseline to 4 weeks is presented here.
Time Frame: baseline and 4 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the FOSQ at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 101 | 103
Units on a scale | 2.2 (0.23) | 1.4 (0.22)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0153, ANCOVA

44. Secondary Outcome: Change From Baseline on Functional Outcomes of Sleep Questionnaire (FOSQ) Total Score at 8 Weeks
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum = 2 maximum = 120) was calculated from the responses. The change in total score from baseline to 8 weeks is presented here.
Time Frame: baseline and 8 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the FOSQ at baseline and at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 97 | 96
Units on a scale | 2.2 (0.25) | 1.4 (0.25)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0296, ANCOVA

45. Secondary Outcome: Change From Baseline on Functional Outcomes of Sleep Questionnaire (FOSQ) Total Score at 12 Weeks
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum = 2 maximum = 120) was calculated from the responses. The change in total score from baseline to 12 weeks is presented here.
Time Frame: baseline and 12 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the FOSQ at baseline and at 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 89 | 93
Units on a scale | 2.6 (0.27) | 1.6 (0.27)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0107, ANCOVA

46. Secondary Outcome: Number of Responders According to the Functional Outcomes of Sleep Questionnaire (FOSQ) Total Score at Endpoint (Week 12 or Last Observation After Baseline)
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum = 2 maximum = 120) was calculated from the responses. A responder analysis defining responders as patients with a total score > 17.9 at Endpoint (12 weeks or last observation after baseline) is presented.
Time Frame: Endpoint (week 12 or last observation after baseline)
Population: Full analysis set defined as subjects with at least one observation after baseline
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 110 | 108
Participants
  Responders | 49 | 30
  Non-responders | 61 | 78
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders are defined as patients with a total score on FOSQ > 17.9; Test type: Superiority or Other; p = 0.0100, Chi-squared — P-value for the treatment comparison is from a Pearson's chi-square test

47. Secondary Outcome: Number of Responders According to the Functional Outcomes of Sleep Questionnaire (FOSQ) Total Score at 2 Weeks
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum=2 maximum=120) was calculated from the responses. A responder analysis defining responders as patients with a total score > 17.9 at 2 weeks is presented here.
Time Frame: 2 weeks following start of study drug administration
Population: Full analysis set defined as subject who completed the FOSQ at 2 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 105 | 103
Participants
  Responders | 30 | 19
  Non-responders | 75 | 84
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders are defined as subjects with a total score of > 17.9; Test type: Superiority or Other; p = 0.0854, Chi-squared — P-value for treatment comparison is from a Pearson's chi-square test

48. Secondary Outcome: Number of Responders According to the Functional Outcomes of Sleep Questionnaire (FOSQ) at Week 4
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum=2 maximum = 120) was calculated from the responses. A responder analysis defining responders as patients with a total score > 17.9 at 4 weeks is presented here.
Time Frame: 4 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the FOSQ at 4 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 105 | 103
Participants
  Responders | 45 | 24
  Non-responders | 60 | 79
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders are defined as subjects with a total score > 17.9; Test type: Superiority or Other; p = 0.0027, Chi-squared — P-value for the treatment comparison is from Pearson's chi-square test

49. Secondary Outcome: Number of Responders According to the Functional Outcomes of Sleep Questionnaire (FOSQ) at Week 8
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score was calculated from the responses (minimum = 2 maximum = 120). A responder analysis defining responders as patients with a total score > 17.9 at 8 weeks is presented here.
Time Frame: 8 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the FOSQ at 8 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 101 | 97
Participants
  Responders | 36 | 20
  Non-responders | 65 | 77
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders are defined as subjects who had a total score of > 17.9; Test type: Superiority or Other; p = 0.0189, Chi-squared — P-value for the treatment comparison is from a Pearson's chi-square test

50. Secondary Outcome: Number of Responders According to the Functional Outcomes of Sleep Questionnaire (FOSQ) at Week 12
Description: The FOSQ is a self-administered questionnaire that assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors. The questionnaire contains 30 questions each rated from 1 to 4 (1 indicating extreme difficulty 4 indicating no difficulty, or 0 indicating not applicable). A total score (minimum = 2 maximum = 120) was calculated from the responses. A responder analysis defining responders as patients with a total score > 17.9 at 12 weeks is presented here.
Time Frame: 12 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who completed the FOSQ at 12 weeks
Measure: Number; unit: Participants
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 94 | 94
Participants
  Responders | 43 | 28
  Non-responders | 51 | 66
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; Responders are defined as subjects with total score > 17.9; Test type: Superiority or Other; p = 0.0240, Chi-squared — P-value for the treatment comparison is from a Pearson's chi-square test

51. Secondary Outcome: Change From Baseline on Medical Outcomes Study 6 Item Cognitive Functioning (MOS-CF6) Scale at Endpoint (12 Weeks or Last Observation After Baseline)
Description: The MOS-CF6 assesses self-reported cognitive function. Items were selected to cover 6 relevant aspects of cognitive functioning:confusion, concentration/thinking, attention, memory, reasoning, problem-solving, and processing speed. Responses range from "none of the time" to "all of the time". The MOS-CF6 is scored by summing responses across the 6 items and converting the total to a 0 - 100 point scale, with the higher score indicating better cognitive functioning. Data is presented showing the change in score from baseline to Endpoint (12 weeks or last observation after baseline).
Time Frame: Baseline and Endpoint (12 weeks or last observation after baseline)
Population: Full analysis set defined as subjects who had at least one observation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 112 | 110
Units on a scale | 3.2 (0.56) | 2.4 (0.56)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.3320, ANCOVA

52. Secondary Outcome: Change From Baseline on Medical Outcomes Study 6 Item Cognitive Functioning (MOS-CF6) Scale at 2 Weeks
Description: The MOS-CF6 assesses self-reported cognitive function. Items were selected to cover 6 relevant aspects of cognitive functioning as follows: confusion, concentration/thinking, attention, memory, reasoning, problem-solving, and processing speed. The MOS-CF6 responses includes 6 choices, ranging from "none of the time" to "all of the time". The MOS-CF6 is scored by summing responses across the 6 items and converting the total to a 0 - 100 point scale, with the higher score indicating better cognitive functioning. Data is presented showing the change in score from baseline to 2 weeks.
Time Frame: baseline and 2 weeks
Population: Full analysis set defined as subjects who completed the MOS-CF6 at baseline and at 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 109 | 104
Units on a scale | 2.0 (0.57) | 1.9 (0.58)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.8930, ANCOVA

53. Secondary Outcome: Change From Baseline on Medical Outcomes Study 6 Item Cognitive Functioning (MOS-CF6) Scale at 4 Weeks
Description: The MOS-CF6 assesses self-reported cognitive function. Items were selected to cover 6 relevant aspects of cognitive functioning as follows: confusion, concentration/thinking, attention, memory, reasoning, problem-solving, and processing speed. The MOS-CF6 responses includes 6 choices, ranging from "none of the time" to "all of the time". The MOS-CF6 is scored by summing responses across the 6 items and converting the total to a 0 - 100 point scale, with the higher score indicating better cognitive functioning. Data is presented showing the change in score from baseline to 4 weeks.
Time Frame: baseline and 4 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the MOS-CF6 at baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 109 | 106
Units on a scale | 3.4 (0.50) | 2.4 (0.51)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.1774, ANCOVA

54. Secondary Outcome: Change From Baseline on Medical Outcomes Study 6 Item Cognitive Functioning (MOS-CF6) Scale at 8 Weeks
Description: The MOS-CF6 assesses self-reported cognitive function. Items were selected to cover 6 relevant aspects of cognitive functioning as follows: confusion, concentration/thinking, attention, memory, reasoning, problem-solving, and processing speed. The MOS-CF6 responses includes 6 choices, ranging from "none of the time" to "all of the time". The MOS-CF6 is scored by summing responses across the 6 items and converting the total to a 0 - 100 point scale, with the higher score indicating better cognitive functioning. Data is presented showing the change in score from baseline to 8 weeks.
Time Frame: baseline and 8 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the MOS-CF6 at baseline and at week 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 104 | 98
Units on a scale | 3.3 (0.49) | 2.1 (0.51)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.1000, ANCOVA

55. Secondary Outcome: Change From Baseline on Medical Outcomes Study 6 Item Cognitive Functioning (MOS-CF6) Scale at 12 Weeks
Description: The MOS-CF6 assesses self-reported cognitive function. Items were selected to cover 6 relevant aspects of cognitive functioning as follows: confusion, concentration/thinking, attention, memory, reasoning, problem-solving, and processing speed. The MOS-CF6 responses includes 6 choices, ranging from "none of the time" to "all of the time". The MOS-CF6 is scored by summing responses across the 6 items and converting the total to a 0 - 100 point scale, with the higher score indicating better cognitive functioning. Data is presented showing the change in score from baseline to 12 weeks.
Time Frame: baseline and 12 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed MOS-CF6 at baseline and at 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 95 | 93
Units on a scale | 3.3 (0.58) | 2.4 (0.59)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.2428, ANCOVA

56. Secondary Outcome: Change From Baseline in the Excessive Sleepiness (ES) Symptom Rating Form - Sleepiness Scores at Endpoint (12 Weeks or Last Observation After Baseline)
Description: The Excessive Sleepiness Symptom Rating Form was used to assess symptoms of excessive sleepiness. Patients rate 7 symptoms(tiredness, fatigue, sleepiness, lack of energy, trouble paying attention, forgetfulness, trouble staying organized) on an 11-point Likert scale (0 = no problem at all to 10 = as bad as you can imagine). ES Symptom Rating Form was designed to follow the response to treatment measuring severity of each of these 7 symptoms using the same 11-point scale. Change from Baseline to Endpoint (12 weeks or last baseline observation) is presented only for the symptom of "Sleepiness".
Time Frame: Baseline and Endpoint (12 weeks or last observation after baseline)
Population: Full analysis set defined as subjects with at least one observation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 112 | 111
Units on a scale | -1.8 (0.24) | -1.4 (0.24)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.1816, ANCOVA

57. Secondary Outcome: Change From Baseline in the Excessive Sleepiness (ES) Symptom Rating Form - Sleepiness Scores at 2 Weeks
Description: Cephalon created the Excessive Sleepiness Symptom Rating Form to assess symptoms of excessive sleepiness. Patients rate 7 symptoms(Tiredness, Fatigue, Sleepiness, Lack of energy, Trouble paying attention, Forgetfulness, Trouble staying organized) each on an 11-point Likert scale(0="no problem at all" 10="as bad as you can imagine"). ES Symptom Rating Form was designed to follow the response to treatment (measuring severity) of each of these 7 symptoms using the same 11-point scale. Change from Baseline to 2 Weeks is presented only for the symptom of "Sleepiness".
Time Frame: Baseline and 2 weeks
Population: Full analysis set defined as subjects who completed the ES Symptom Rating form at baseline and 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 106 | 105
Units on a scale | -1.6 (0.22) | -1.2 (0.22)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.1627, ANCOVA

58. Secondary Outcome: Change From Baseline in the Excessive Sleepiness (ES) Symptom Rating Form - Sleepiness Scores at 4 Weeks
Description: Cephalon created the Excessive Sleepiness Symptom Rating Form to assess symptoms of excessive sleepiness. Patients rate 7 symptoms(Tiredness, Fatigue, Sleepiness, Lack of energy, Trouble paying attention, Forgetfulness, Trouble staying organized) each on an 11-point Likert scale(0="no problem at all" 10="as bad as you can imagine"). ES Symptom Rating Form was designed to follow the response to treatment (measuring severity) of each of these 7 symptoms using the same 11-point scale. Change from Baseline to 4 Weeks is presented only for the symptom of "Sleepiness".
Time Frame: Baseline and 4 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the ES Symptom Rating Form at Baseline and at 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 110 | 106
Units on a scale | -2.1 (0.23) | -1.1 (0.23)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0018, ANCOVA

59. Secondary Outcome: Change From Baseline in the Excessive Sleepiness (ES) Symptom Rating Form - Sleepiness Scores at 8 Weeks
Description: Cephalon created the Excessive Sleepiness Symptom Rating Form to assess symptoms of excessive sleepiness. Patients rate 7 symptoms(Tiredness, Fatigue, Sleepiness, Lack of energy, Trouble paying attention, Forgetfulness, Trouble staying organized) each on an 11-point Likert scale(0="no problem at all" 10="as bad as you can imagine"). ES Symptom Rating Form was designed to follow the response to treatment (measuring severity) of each of these 7 symptoms using the same 11-point scale. Change from Baseline to 8 Weeks is presented only for the symptom of "Sleepiness".
Time Frame: baseline and 8 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the ES Symptom Rating Form at baseline and at 8 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 103 | 98
Units on a scale | -1.8 (0.24) | -0.9 (0.25)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0096, ANCOVA

60. Secondary Outcome: Change From Baseline in the Excessive Sleepiness (ES) Symptom Rating Form - Sleepiness Scores at 12 Weeks
Description: Cephalon created the Excessive Sleepiness Symptom Rating Form to assess symptoms of excessive sleepiness. Patients rate 7 symptoms(Tiredness, Fatigue, Sleepiness, Lack of energy, Trouble paying attention, Forgetfulness, Trouble staying organized) each on an 11-point Likert scale(0="no problem at all" 10="as bad as you can imagine"). ES Symptom Rating Form was designed to follow the response to treatment (measuring severity) of each of these 7 symptoms using the same 11-point scale. Change from Baseline to 12 Weeks is presented only for the symptom of "Sleepiness".
Time Frame: Baseline and 12 weeks following start of study drug administration
Population: Full analysis set defined as subjects who completed the ES Symptom Rating Form at baseline and at 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 95 | 94
Units on a scale | -2.2 (0.25) | -1.3 (0.25)
Statistical Analysis 1: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0126, ANCOVA

ADVERSE EVENTS:
Arm/Group | Armodafinil 200 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/124 | 3/124
Other Adverse Events (participants affected / at risk) | 56/124 | 34/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 200 mg/Day (N=124) | Placebo (N=124)
Angina unstable (Cardiac disorders) | 0 (0) | 1
Chest pain (General disorders) | 1 | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 200 mg/Day (N=124) | Placebo (N=124)
Dry Mouth (Gastrointestinal disorders) | 10 | 0
Nausea (Gastrointestinal disorders) | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Irritability (General disorders) | 5 | 1
Feeling jittery (General disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 7
Nasopharyngitis (Infections and infestations) | 5 | 6
Headache (Nervous system disorders) | 14 | 9
Dizziness (Nervous system disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 9 | 2
Anxiety (Psychiatric disorders) | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days